CLINICAL TRIAL: NCT03447249
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Brief Title: A Phase 3 Study of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VX17-659-102; 2017-004132-11 (EudraCT Number)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants who received placebo matched to VX-659/TEZ/IVA for 24 weeks in the TC treatment period.
  Interventions: Drug: Placebo
- VX-659/TEZ/IVA TC (Experimental): Participants who received VX-659 240 mg/TEZ 100 mg/IVA 150 mg as fixed-dose combination (FDC) tablets in the morning and IVA 150 mg as mono tablet in the evening for 24 weeks in the TC treatment period.
  Interventions: Drug: VX-659/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: VX-659/TEZ/IVA — Participants received VX-659/TEZ/IVA orally once daily in the morning.
  Other Names: VX-659/VX-661/VX-770; VX-659/tezacaftor/ivacaftor
  Arms: VX-659/TEZ/IVA TC
Drug: IVA — Participants received IVA orally once daily in the evening.
  Other Names: VX-770; ivacaftor
  Arms: VX-659/TEZ/IVA TC
Drug: Placebo — Participants received placebo matched VX-659/TEZ/IVA orally once daily in the morning and placebo matched to IVA orally once daily in the evening.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of VX-659 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are heterozygous for F508del and a minimal function mutation (F/MF subjects).

ELIGIBILITY:
Key Inclusion Criteria:

* Heterozygous for F508del and an MF mutation (as defined in the protocol)
* Forced expiratory volume in 1 second (FEV1) value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (101):
- United States (48):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Hartford Health, Hartford, Connecticut
  - Yale New Haven Medical Center, New Haven, Connecticut
  - University of Miami/ Miller School of Medicine, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - Advocate Children's Hospital - Park Ridge/ North Suburban Pulmonary and Critical Care Consultants, Niles, Illinois
  - Indiana Clinical Research Center, IU Health University Hospital, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kentucky Clinic, Lexington, Kentucky
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital CF Center, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine/ St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, Lebanon, New Hampshire
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - Lung and Cystic Fibrosis Center at Women and Children's Hospital of Buffalo, Buffalo, New York
  - Northwell Health, Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Respiratory Diseases of Children and Adolescents, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Drexel University College of Medicine/ Drexel Adult Cystic Fibrosis Center, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Research/ USD, Sioux Falls, South Dakota
  - University of Tennessee Medical Center - Adult Cystic Fibrosis Clinic, Knoxville, Tennessee
  - Children's Foundation Research Center/ Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Pediatric Pulmonary & Allergy/Immunology Clinic, Spokane, Washington
- Australia (8):
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Chermside
  - Royal Brisbane & Women's Hospital, Herston
  - Institute for Respiratory Health Inc./ Sir Charles Gairdner Hospital, Nedlands
  - John Hunter Hospital & Hunter Medical Research Institute, New Lambton Heights
  - Sydney Children's Hospital, Randwick, Randwick
  - Princess Margaret Hospital for Children, Subiaco
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- Germany (9):
  - Charite Paediatric Pulmonology Department, Berlin
  - University Hospital Cologne, Cologne
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Clinic of J.W Goethe University, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Mukeviszidose-Zentrum am Universitatsklinikum Jena, Klinik fuer Kinder - und Jugendmedizin, Jena
  - Universitatsklinikum Schleswig-Holstein, Klinik fur Kinder- und Jugendmedizin, Lübeck
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologische Praxis Pasing, München
- Ireland (7):
  - Beaumont Hospital, Dublin
  - Children's University Hospital Temple Street, Dublin
  - Cork University Hospital, Dublin
  - Our Lady's Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - National University of Ireland, Galway
  - University Hospital Limerick, Limerick
- Israel (5):
  - Lady Davis Carmel Medical Center, Haifa
  - Pediatric Pulmonary Unit Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Instytut Matki i Dziecka, Warsaw, Poland
- Spain (7):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d'Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infantil La Paz, Madrid
  - Coporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Switzerland (3):
  - Lindenhofspital - Quartier Bleu, Bern
  - Kinderspital Zuerich, Zurich
  - Universitaetsspital Zuerich, Zurich
- United Kingdom (9):
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Queen Elizabeth University Hospital, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Queens Medical Center, Nottingham
  - University Hospital Llandough, Penarth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 385 participants were enrolled in the study, of which 3 participants were enrolled but were not dosed in the TC treatment period. Results are presented for 382 participants dosed in the TC treatment period.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 12 years or older.
Groups:
- Placebo: Participants who received placebo matched to VX-659/TEZ/IVA in the morning and placebo matched to IVA in the evening for 24 weeks in the TC treatment period.
Period: Overall Study
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Started | 190 | 192
Safety Set (Based on actual treatment received.) | 189 | 193
Completed | 185 | 192
Not Completed | 5 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal of consent (not due to AE) | 1 | 0
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who carried the intended CF transmembrane conductance regulator gene (CFTR) allele mutation and received at least 1 dose of study drug in the TC Treatment Period.
Groups:
- VX-659/TEZ/IVA TC: Participants who received VX-659 240 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA 150 mg as mono tablet in the evening for 24 weeks in the TC treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-659/TEZ/IVA TC | Total
Number analyzed (Participants) | 190 | 192 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (10.0) | 26.7 (9.8) | 26.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 168
  Male | 107 | 107 | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 181 | 184 | 365
  Unknown or Not Reported | 2 | 2 | 4
Race [Count of Participants; unit: Participants]
  White | 187 | 188 | 375
  Black or African American | 1 | 2 | 3
  Both White and Black/African American | 2 | 2 | 4
Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percentage points | 60.4 (14.5) | 60.7 (15.4) | 60.6 (14.9)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Week 4
Population: Analysis population included all participants in the Full Analysis Set (all randomized participants who carried the intended CFTR allele mutation and received at least 1 dose of study drug) who completed the Week 4 Visit or were randomized at least 28 days before the data cutoff date.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
percentage points | -1.0 (0.6) | 13.0 (0.6)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; The data presented for Primary endpoint was based on interim analysis at Week 4; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; Least Squares (LS) Mean Difference = 14.0, 95% CI 2-sided [12.4 to 15.7]

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Week 24
Population: Full analysis set (FAS) included all randomized participants who carried the intended CFTR allele mutation and received at least 1 dose of study drug in the TC Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
percentage points | -0.8 (0.6) | 13.4 (0.6)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 14.2, 95% CI 2-sided [12.6 to 15.7]

3. Secondary Outcome: Number of Pulmonary Exacerbations (PEx)
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Number; unit: pulmonary exacerbation events
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
pulmonary exacerbation events | 116 | 17
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Negative binomial regression model; Rate ratio = 0.14, 95% CI 2-sided [0.09 to 0.24]

4. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
millimole per liter (mmol/L) | -0.1 (1.0) | -44.6 (0.9)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = -44.6, 95% CI 2-sided [-47.2 to -41.9]

5. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
units on a scale | -1.5 (1.1) | 18.6 (1.0)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 20.1, 95% CI 2-sided [17.2 to 23.0]

6. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: From Baseline at Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: kilogram per meter square (kg/m^2)
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
kilogram per meter square (kg/m^2) | -0.05 (0.07) | 1.06 (0.07)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 1.11, 95% CI 2-sided [0.91 to 1.31]

7. Secondary Outcome: Absolute Change in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
mmol/L | 0.0 (1.0) | -43.3 (1.0)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = -43.4, 95% CI 2-sided [-46.3 to -40.5]

8. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) Respiratory Domain Score
Description: as for outcome 5
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
units on a scale | 0.1 (1.2) | 18.0 (1.2)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 17.9, 95% CI 2-sided [14.5 to 21.3]

9. Secondary Outcome: Time-to-first Pulmonary Exacerbation (PEx)
Description: as for outcome 3
Time Frame: From Baseline through Week 24
Population: FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
days | NA [NA to NA] — Median and 95% confidence interval could not be estimated because less than 50% of participants had events. | NA [NA to NA] — Median and 95% confidence interval could not be estimated because less than 50% of participants had events.

10. Secondary Outcome: Absolute Change in BMI Z-score for Participants <=20 Years of Age at Baseline
Description: BMI was defined as weight in kg divided by height in m^2. z-score is a statistical measure to describe whether a mean was above or below the standard. BMI, adjusted for age and sex, was analyzed as BMI-for-age z-score. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI.
Time Frame: From Baseline at Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were <=20 years of age at Baseline.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 59 | 58
kg/m^2 | -0.08 (0.05) | 0.31 (0.05)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; LS Mean Difference = 0.39, 95% CI 2-sided [0.24 to 0.54]

11. Secondary Outcome: Absolute Change in Body Weight
Time Frame: From Baseline at Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 190 | 192
kg | 0.1 (0.2) | 3.3 (0.2)
Statistical Analysis 1: Comparison: Placebo vs VX-659/TEZ/IVA TC; Test type: Superiority; LS Mean Difference = 3.2, 95% CI 2-sided [2.7 to 3.8]

12. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to 28 weeks)
Population: Adverse events are presented as per Safety Set. Group assignments for participants in the Safety Set were based on actual treatment received, such that 1 participant assigned to Placebo group who inadvertently received one or more doses of VX-659/TEZ/IVA TC regimen was included in VX-659/TEZ/IVA TC group for the purpose of safety analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 189 | 193
participants
  Participants with TEAEs | 175 | 173
  Participants with Serious TEAEs | 58 | 11

13. Secondary Outcome: Observed Pre-dose Concentration (Ctrough) of VX-659, TEZ, M1-TEZ, and IVA
Time Frame: Pre-dose on Week 4, 8, 12, and 16
Population: Pharmacokinetic (PK) set included all randomized participants who carried the intended CFTR allele mutation and received at least 1 dose of study drug in the TC Treatment Period. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 192
nanogram per milliliter (ng/mL)
  VX-659 (Week 4): number analyzed (Participants) | 150
  VX-659 (Week 4) | 662 (528)
  VX-659 (Week 8): number analyzed (Participants) | 148
  VX-659 (Week 8) | 764 (1520)
  VX-659 (Week 12): number analyzed (Participants) | 144
  VX-659 (Week 12) | 614 (519)
  VX-659 (Week 16): number analyzed (Participants) | 162
  VX-659 (Week 16) | 638 (521)
  TEZ (Week 4): number analyzed (Participants) | 150
  TEZ (Week 4) | 1220 (645)
  TEZ (Week 8): number analyzed (Participants) | 148
  TEZ (Week 8) | 1390 (1250)
  TEZ (Week 12): number analyzed (Participants) | 142
  TEZ (Week 12) | 1290 (766)
  TEZ (Week 16): number analyzed (Participants) | 161
  TEZ (Week 16) | 1220 (654)
  M1-TEZ (Week 4): number analyzed (Participants) | 150
  M1-TEZ (Week 4) | 4380 (1560)
  M1-TEZ (Week 8): number analyzed (Participants) | 148
  M1-TEZ (Week 8) | 4580 (1480)
  M1-TEZ (Week 12): number analyzed (Participants) | 142
  M1-TEZ (Week 12) | 4580 (1530)
  M1-TEZ (Week 16): number analyzed (Participants) | 161
  M1-TEZ (Week 16) | 4420 (1520)
  IVA (Week 4): number analyzed (Participants) | 150
  IVA (Week 4) | 442 (277)
  IVA (Week 8): number analyzed (Participants) | 148
  IVA (Week 8) | 548 (1100)
  IVA (Week 12): number analyzed (Participants) | 142
  IVA (Week 12) | 429 (327)
  IVA (Week 16): number analyzed (Participants) | 161
  IVA (Week 16) | 416 (303)

ADVERSE EVENTS:
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to 28 weeks)
Description: Adverse events are presented as per Safety Set. Group assignments for participants in the Safety Set were based on actual treatment received, such that 1 participant assigned to Placebo group who inadvertently received one or more doses of VX-659/TEZ/IVA TC regimen was included in VX-659/TEZ/IVA TC group for the purpose of safety analysis.
Arm/Group | Placebo | VX-659/TEZ/IVA TC
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/193
Serious Adverse Events (participants affected / at risk) | 58/189 | 11/193
Other Adverse Events (participants affected / at risk) | 166/189 | 141/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=189) | VX-659/TEZ/IVA TC (N=193)
Intentional self-injury (Psychiatric disorders) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 0 | 1
Right-to-left cardiac shunt (Congenital, familial and genetic disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Device damage (Product Issues) | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 45 | 3
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Dysentery (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=189) | VX-659/TEZ/IVA TC (N=193)
Alanine aminotransferase increased (Investigations) | 2 | 17
Blood creatine phosphokinase increased (Investigations) | 7 | 13
Aspartate aminotransferase increased (Investigations) | 4 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 68 | 34
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 38 | 28
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 | 6
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 14 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Headache (Nervous system disorders) | 31 | 26
Pyrexia (General disorders) | 15 | 13
Fatigue (General disorders) | 19 | 9
Diarrhoea (Gastrointestinal disorders) | 16 | 17
Nausea (Gastrointestinal disorders) | 24 | 8
Abdominal pain upper (Gastrointestinal disorders) | 10 | 3
Vomiting (Gastrointestinal disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 5 | 11
Rash (Skin and subcutaneous tissue disorders) | 10 | 10
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 79 | 21
Upper respiratory tract infection (Infections and infestations) | 7 | 35
Nasopharyngitis (Infections and infestations) | 16 | 26
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT03447249/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03447249/SAP_001.pdf